CLINICAL TRIAL: NCT04731506
Title: Family Connections: Cultural Adaptation and Feasibility Testing of a Technology-based Pediatric Weight Management Intervention for Rural Latino Communities
Brief Title: Family Connections: Cultural Adaptation and Feasibility Testing for Rural Latino Communities
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator returned to home country for cancer treatment.
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); University of Nebraska Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0745-20-EP; P20GM104320 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-05

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Experimental): Parent participants will receive an activity workbook that promotes increased physical activity, healthy diets and decreased screen time, two in-person support sessions spaced and 10 Interactive Voice Response (IVR) automated telephone system calls providing health education messages over 12 months.
  Participants in the "standard care" arm include parent-child dyads. Data are collected from both parents and their children; however, only parents participate in intervention activities (workbook, classes, calls).
  Interventions: Behavioral: Family Connections
- Waitlist (No Intervention): Participants randomized into the control group will receive an activity workbook that promotes increased physical activity, healthy diets, and decreased screen time. They will be waitlisted (placed on a 6-month delayed start) to receive the full Family Connections program.
  Participants in the "waitlist" arm include parent-child dyads. Data are collected from both parents and their children; however, only parents later participate in intervention activities (workbook, classes, calls).

INTERVENTIONS:
Behavioral: Family Connections — Parent participants will receive an activity workbook that promotes increased physical activity and consumption of fruits and vegetables and decreased screen time and intake of sugary drink consumption, two in-person support sessions to help parents to develop an action plan spaced one week apart & Interactive Voice Response (IVR) automated telephone system calls of 5 to 10 minutes that provide health education messages over 12 months (4 weekly, 4 biweekly (4), and 2 monthly). During each IVR call parents provide information on current physical activities, and food consumption that is used to provide feedback on success in subsequent IVR calls.
  Arms: Standard Care

SUMMARY:
There are marked ethnic and rural-urban disparities in the prevalence of childhood obesity (CO). Among Latino/Hispanic children, CO is almost 60% higher than that of non- Latino/Hispanic Whites, and among children in rural areas it is estimated to be 25% to almost 50% higher that of urban areas. By 2050 Latinos are expected to represent 51.2% of rural Nebraska's population, so addressing childhood obesity risk factors among Latinos/Hispanic families living in rural communities and Identifying effective interventions is an important priority. The first aim will be to collaboratively adapt all intervention materials to better fit the rural Latino/Hispanic community, including translation of materials to Spanish, inclusion of culturally relevant content and images, and use of health communication strategies to address different levels of health literacy. The second aim randomly assign enrolled participant dyads (parent and child) to either Family Connections (FC) or a waitlist standard-care (SC) group to determine preliminary effectiveness in reducing child body mass index (BMI) z-score (a standardized way to measure a child's weight in relation to their age and sex). This study will address three important questions as they apply to Latino/Hispanic in rural Nebraska: is a telephone delivered family-based childhood obesity (FBCO) program in rural Nebraska culturally relevant, usable and acceptable, is a telephone delivered FBCO program effective at reducing child BMI z-scores and what real-world factors influence the impact of the intervention to sustainably engage a meaningful population of Latino/Hispanic families who stand to benefit.

DETAILED DESCRIPTION:
The childhood obesity (CO) rate of Latinos/Hispanics, the fastest growing rural population group, is 60% higher than their non-Hispanic neighbors. Family-based childhood obesity (FBCO) interventions targeting parents have shown promising results for reducing weight among children. However, these interventions are developed and evaluated with culturally homogeneous samples of participants in large urban areas and have been poorly accessed by Latino/Hispanic families living in rural communities. There are a number of barriers to accessing these interventions in rural Nebraska communities including increasing ethnic health disparities, limited available resources, shortage of available health professionals, and the existence of demographically and geographically segregated communities. Community members have reported that family and work responsibilities, lack of public transportation, and language and cultural relevance have kept them from engaging in these programs. Interactive technologies may provide a possible solution to these challenges in that they offer an avenue for the delivery of FBCO interventions at times and places convenient to participants.

Investigators have found that a technology-assisted FBCO intervention can lead to significant weight loss among children and that over 82% of Latinos/Hispanics in studies have mobile devices regularly used to access information and make phone calls. Thus, telephone systems that provide automated (i.e., interactive voice response (IVR) system) FBCO messages may be practical methods for delivering culturally appropriate health information and engaging Latino/Hispanic families in rural communities. Family Connections (FC) is a scalable intervention that uses IVR to deliver FBCO content; however, it was not specifically developed for Latino/Hispanic rural families.

This study will build on investigators' experience in the use of interactive technologies to deliver FBCO content and promote healthy behaviors and weight control, culturally adapting interventions and working collaboratively with stakeholders in a variety of settings. The first aim is to culturally adapt a relevant and acceptable technology-delivered FBCO intervention. A mixed-methods approach will be used that includes a community workgroup facilitated by our rural partner organizations in Nebraska and a using structured community input adaptation process. The next study aim will follow-up to evaluate the feasibility and preliminary effectiveness of this intervention with Latino/Hispanic rural families in Nebraska. Participants will be randomly assigned to one of two groups: a technology-delivered Family Connections (FC) group or a waitlist standard-care (SC) group. Both groups will receive a workbook. The FC group will additionally receive two in-person group sessions followed by 10 IVR calls over a period of 12 months. The two groups will be compared to determine program effectiveness in reducing child BMI z-scores, diet, physical activity, health literacy, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Intervention Adult Participants

* Age ≥ 19 years
* Self-identified as Latino/Hispanic living in target counties
* Parent of a child aged 8-12 years with a BMI z-score ≥85th
* Willing and able to give informed consent

Children Participants

* Age 6-12 years
* Body Mass Index (BMI) z-score ≥85th percentile
* Self-Identified as Latino/Hispanic living in target counties
* Assent to participate in the study

Exclusion Criteria:

* Contraindication to physical activity or weight loss
* Planning to move in the next 12 months
* Currently participating in weight loss program
* Pregnancy or planning to get pregnant in the next 12 months
* Not willing to be randomized
* Not willing to consent or assent to participate

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tzeyu Michaud, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Summary results will be shared with all identifiers removed at the completion of the study after all analyses have been finalized.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Summary results (de-identified) will be shared at the completion of the study.
Access Criteria: Request submitted to the to the Principal Investigator.

REFERENCES:
- [Derived] Brito FA, Alves TF, Santos N, Michaud TL, Eisenhauer C, De Leon EB, Squarcini CFR, Kachman S, Almeida F, Estabrooks P. Feasibility of a culturally adapted technology-delivered, family-based childhood obesity intervention for Latino/Hispanic families in rural Nebraska: the Hispanic Family Connections study protocol. BMJ Open. 2024 Oct 18;14(10):e089186. doi: 10.1136/bmjopen-2024-089186. PMID 39424377

RESULTS

PARTICIPANT FLOW:
Groups:
- Parent- Standard Care: Parent participants will receive an activity workbook that promotes increased physical activity, healthy diets, and decreased screen time, two in-person support sessions spaced, and 10 Interactive Voice Response (IVR) automated telephone system calls providing health education messages over 12 months.
- Parent- Waitlist: Parent participants who are wait-listed will receive an activity workbook that promotes increased physical activity, healthy diets, and decreased screen time, and then will be placed on a 6-month delayed start (wait-list) in the FC program.
- Child- Standard Care: Children directly participated in data collection at baseline and 12 months. Children did not participate in the intervention activities led by the research team. Their parents (parent- standard care) received an activity workbook that promotes increased physical activity, healthy diets and decreased screen time, two in-person support sessions, and 10 Interactive Voice Response (IVR) automated telephone system calls providing health education messages over 12 months.
- Child- Waitlist: Children directly participated in data collection at baseline and 12 months. Children did not participate in the intervention activities led by the research team. Their parents (parent- wait-list) were wait-listed and received an activity workbook that promotes increased physical activity, healthy diets, and decreased screen time. Then they were placed on a 6-month wait-list (delayed start) in the FC program.
Period: Overall Study
Arm/Group | Parent- Standard Care | Parent- Waitlist | Child- Standard Care | Child- Waitlist
Started | 25 | 13 | 26 | 12
Completed | 8 | 11 | 8 | 10
Not Completed | 17 | 2 | 18 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parent- Standard Care | Child- Standard Care | Parent- Waitlist | Child- Waitlist | Total
Number analyzed (Participants) | 25 | 26 | 13 | 12 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (1.6) | 9.8 (2.2) | 37.2 (9.5) | 9.8 (8.2) | 24.05 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 24 | 13 | 7 | 58
  Male | 11 | 2 | 0 | 5 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Z-score [Mean (Standard Deviation); unit: z-score] — BMI z-score is a measurement for children Population: Z-score for children only
  z-score
    number analyzed (Participants) | 0 | 26 | 0 | 12 | 38
    (all) |  | 2.1 (0.4) |  | 1.7 (0.8) | 2.0 (0.6)
BMI [Mean (Standard Deviation); unit: Kg/m^2] — BMI is a measurement for adults Population: BMI for adults
  Kg/m^2
    number analyzed (Participants) | 25 | 0 | 13 | 0 | 38
    (all) | 32.2 (6.3) |  | 37.7 (13.9) |  | 34.1 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Child- Change in BMI Z-score at 12 Months From Baseline
Description: We used the mixed-effect regression model for the BMI z-score, weight, and BMI, regardless adults or kids. Weight was measured with a calibrated Heavy-Duty digital floor scale 880KL (www.homscales.com) in stocking feet. For a child's BMI z-score, we use the formula Z=((BMI/M)^{L}-1)/(L\times S), where M, L, and S are parameters specific to the child's sex and age. For specific age and sex combinations, the parameters M, L, and S are obtained from reference data tables, provided by the CDC (https://www.cdc.gov/growthcharts/extended-bmi-data-files.htm). A Z-score indicates how many standard deviations a data point is from the mean.
  For children and adolescents, specific z-score ranges are used to define weight status: (Negative Z-score, below mean) underweight (<-2), healthy weight (-2 to +1), (Positive Z-score, above mean) overweight (+1 to +2), and obese (>+2).
  Z-scores & Health: ≥0 greater risk for developing cardiovascular disease. <-2 osteoporosis and bone fractures risk.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: BMI z score (children)
Groups:
- Child- Waitlist: Children directly participated in data collection at baseline and 12 months. Children did not participate in the intervention activities led by the research team. Their parents (parent- waitlist) were waitlisted and received an activity workbook that promotes increased physical activity, healthy diets, and decreased screen time. Then they were placed on a 6-month waitlist (delayed start) in the FC program.
Arm/Group | Child- Standard Care | Child- Waitlist
Number analyzed (Participants) | 8 | 10
BMI z score (children) | -0.158 (0.133) | -0.031 (0.276)
Statistical Analysis 1: Comparison: Child- Waitlist; BMI z-score analysis is for children only; Test type: Superiority; p = 0.286, Mann-Whitney U test — Difference between Child-standard care and Child-waitlist arms of respective changes from baseline to 12 months with each arm; We used the Mann-Whitney U test to asses the difference in BMI z-score by arms for child; Mean Difference (Net) = -0.127, 95% CI 2-sided [-0.353 to 0.099]

2. Primary Outcome: Adult- Change in BMI at 12 Months From Baseline
Description: Adult participant's Body Mass Index (BMI), a standardized way to measure an adult's weight in relation to their height, will be determined at the initial in-person visit, then again at 12 months. Height will be measured in stocking feet with a calibrated stadiometer with a fixed vertical backboard and adjustable headboard. Weight will be measured with a calibrated Heavy-Duty digital floor scale 880KL (www.homscales.com) in stocking feet. BMI will be calculated in kg/m2 using the established Centers for Disease Control and Prevention protocol. Higher scores mean a worse outcome. Comparisons of scores at the time points will be made between groups to evaluate program effectiveness.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: BMI = kg/m²
Groups:
- Parent- Waitlist: Parent participants who are waitlisted will receive an activity workbook that promotes increased physical activity, healthy diets, and decreased screen time, and then will be placed on a 6-month delayed start (waitlist) in the FC program.
Arm/Group | Parent- Standard Care | Parent- Waitlist
Number analyzed (Participants) | 8 | 11
BMI = kg/m² | -0.700 (3.14) | -4.35 (12.49)
Statistical Analysis 1: Comparison: Parent- Standard Care vs Parent- Waitlist; Test type: Superiority; p = 0.741, Mann-Whitney U test; We used the Mann-Whitney U test to examine the BMI difference between arms at 12 months for adults; Mean Difference (Net) = 3.65, 95% CI 2-sided [-5.95 to 13.26]

ADVERSE EVENTS:
Time Frame: 12 months.
Description: All-Cause Mortality, Serious, or other (non-serious) Adverse Events were monitored and assessed. The protocol states, "An assessment of potential adverse events will be used to document potential problems and if those problems were related to participation in the program… The study will be audited beginning six months after the start of participant accrual and then annually.
Groups:
- Parent/Child Dyad- Standard Care: Children directly participated in data collection at baseline and 12 months. Children did not participate in the intervention activities led by the research team. Their parents (parent- standard care) received an activity workbook that promotes increased physical activity, healthy diets and decreased screen time, two in-person support sessions, and 10 Interactive Voice Response (IVR) automated telephone system calls providing health education messages over 12 months.
- Parent/Child- Waitlist: Children directly participated in data collection at baseline and 12 months. Children did not participate in the intervention activities led by the research team. Their parents (parent- waitlist) were waitlisted and received an activity workbook that promotes increased physical activity, healthy diets, and decreased screen time. Then they were placed on a 6-month waitlist (delayed start) in the FC program.
Arm/Group | Parent/Child Dyad- Standard Care | Parent/Child- Waitlist
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/25
Other Adverse Events (participants affected / at risk) | 0/51 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT04731506/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Form_English (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT04731506/ICF_001.pdf
  • Informed Consent Form: Informed Consent Form_Spanish (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT04731506/ICF_002.pdf